CLINICAL TRIAL: NCT07297940
Title: An Open Label, Randomized, Single Dose, 2-sequence, 2-period, Cross-over Study to Evaluate the Pharmacokinetics and Safety of DA-1229_01 in Healthy Subjects at Fasting State
Brief Title: Pharmacokinetics and Safety Profiles of DA-1229_01 in Healthy Subjects at Fasting State
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA1229_01-M_Fast_BE
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental)
  Interventions: Drug: DA-1229_01; Drug: DA-1229_01-R
- Sequence B (Experimental)
  Interventions: Drug: DA-1229_01; Drug: DA-1229_01-R

INTERVENTIONS:
Drug: DA-1229_01 — single dose administration (DA-1229 one tablet once a day)
Drug: DA-1229_01-R — single dose administration (DA-1229_01-R one tablet once a day)

SUMMARY:
This clinical study is to evaluate the safety/tolerability and pharmacokinetics of DA-1229_01 at fasting state.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* BMI between 18 and 30 kg/m2
* Body weight: Male ≥ 50kg, Female ≥ 45kg
* Subjects who have signed an informed consent themselves after receiving detailed explanation about clinical study

Exclusion Criteria:

* Subjects with clinically significant medical history
* Subjects with history of drug abuse or addicted
* Subjects with allergy or drug hypersensitivity

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
AUCt | pre-dose~72 hours post-dose
  Area Under the Curve
Cmax | pre-dose~72 hours post-dose
  Maximum Plasma Concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Bumin hospital, Seoul, South Korea